CLINICAL TRIAL: NCT02191098
Title: Proof of Principle Study of Pulse Dosing of IL-15 to Deplete the Reservoir in HIV Infected People on Optimized ART With Undetectable Plasma HIV RNA
Brief Title: Proof of Principle Study of Pulse Dosing of IL-15 to Deplete the Reservoir in HIV Infected People
Acronym: ALT-803
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1508M77601-1
Record Dates: First submitted 2014-07-08; First posted 2014-07-16 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: HIV; Stable ART
Keywords: HIV; ART
MeSH Terms: interventions — ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALT-803 (Experimental): ALT-803
  Interventions: Drug: ALT-803

INTERVENTIONS:
Drug: ALT-803 — Interleukin 15 (IL-15) is a common γ-chain cytokine that is related to interleukin-2 (IL-2) and is a critical factor for the development, proliferation, and activation of effector natural killer (NK) and CD8+ memory T cells

SUMMARY:
To assess the safety and tolerability of ALT-803, as well as, the potential efficacy of ALT-803 in HIV

DETAILED DESCRIPTION:
This is an open-label, single-arm intra-patient dose escalating pilot study of ALT-803, a recombinant human super agonist interleukin-15 (IL-15) complex with an expansion cohort at the maximum tolerated dose (MTD). The primary aim is to investigate the safety and tolerability of ALT-803 in HIV-infected people receiving potent and optimized antiretroviral therapy. All infusions will occur on a Monday. Subjects will be monitored for 24 hours after the first infusion and then for 6 hours after each subsequent infusion, provided no unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected adults aged 18 years or over.
2. Stable ART for at least 36 months
3. Screening plasma HIV RNA levels below level of quantification (<40 to <50 copies RNA/mL depending on the assay) ≥ 2 years (a single measurement above the level of detection but < 100-200 copies/ml will be allowed)
4. Screening CD4 count ≥500 cells/mm3
5. Laboratory tests performed within 14 days of study enrollment:

   1. WBC ≥ 3000/mm3
   2. Platelets ≥ 50,000/mm3 [Patients may be transfused to meet this requirement]
   3. Hemoglobin ≥ 8 g/dL (>80g/L) [Patients may be transfused to meet this requirement]
   4. Calculated glomerular filtration rate (GFR) >45 mL/min/1.73m2
   5. Total bilirubin ≤ 2.0 X upper limit of institutional normal (ULN)
   6. AST, ALT, ALP ≤ 2.0 X ULN
6. Adequate pulmonary function without any clinical sign of severe pulmonary dysfunction. PFTs > 50% of predicted if symptomatic or prior known impairment.
7. Ability to be off prednisone and other immunosuppressive drugs for at least 14 days before first dose of study drug
8. Women of child bearing potential and men with partners of child bearing potential must agree to use effective contraception during therapy and for 4 months after completion of therapy
9. Voluntary written consent

Exclusion Criteria:

1. Active infection other than HIV currently requiring systemic antimicrobial therapy
2. Previously treated on this study or received previous ALT-803
3. Latent TB infection or active TB disease prior to completing a standard regimen of anti-TB therapy
4. Active fungal infection requiring systemic antifungal therapy
5. Active or recurrent herpes or varicella-zoster virus infection requiring treatment (or chronic suppression)
6. Chronic hepatitis B or C
7. Planning or current pregnancy or breastfeeding
8. Intended modification of antiretroviral therapy in the next 24 weeks
9. NYHA (New York Heart Association) Class III or IV heart failure, uncontrollable supraventricular arrhythmias, any history of a ventricular arrhythmia, or other clinical signs of severe cardiac dysfunction
10. Symptomatic congestive heart failure, unstable angina pectoris, or Myocardial infarction within 6 months prior to screening
11. Marked baseline prolongation of QT/QTc interval (e.g. demonstration of a QTc interval greater than 500 milliseconds)
12. History or evidence of uncontrollable CNS disease
13. Prior organ allograft or allogeneic transplantation
14. On-going chronic systemic or regular inhaled corticosteroid use or other immunosuppressive therapy (a history of mild asthma not requiring therapy is eligible)
15. Psychiatric illness/social situations that would limit compliance with study requirements
16. Other illness that in the opinion of the investigator would exclude the patient from participating in this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of ALT-803 in HIV-infected subjects | 4 weeks
  Safety and tolerability is determined by the incidence of adverse events, size of the inducible reservoir as estimated using the TILDA assay

SECONDARY OUTCOMES:
Assess the impact of ALT-803 on the size of the inducible reservoir, | 4 weeks
  Assess the impact of ALT-803 on the size of the inducible reservoir, as estimated using the TILDA assay, in total CD4+ T cells and memory subsets

CONTACTS AND LOCATIONS:
Overall Officials: Tim Schacker, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Miller JS, Davis ZB, Helgeson E, Reilly C, Thorkelson A, Anderson J, Lima NS, Jorstad S, Hart GT, Lee JH, Safrit JT, Wong H, Cooley S, Gharu L, Chung H, Soon-Shiong P, Dobrowolski C, Fletcher CV, Karn J, Douek DC, Schacker TW. Safety and virologic impact of the IL-15 superagonist N-803 in people living with HIV: a phase 1 trial. Nat Med. 2022 Feb;28(2):392-400. doi: 10.1038/s41591-021-01651-9. Epub 2022 Jan 31. PMID 35102335